CLINICAL TRIAL: NCT00762255
Title: A Phase I Trial of Vorinostat in Combination With Bevacizumab and Irinotecan in Recurrent Glioblastoma
Brief Title: A Phase I Trial of Vorinostat in Combination With Bevacizumab & Irinotecan in Recurrent Glioblastoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-15629; 33726 (Other: Merck & Co., Inc.)
Record Dates: First submitted 2008-09-29; First posted 2008-09-30 (Estimated); Last update posted 2013-07-25 (Estimated); Status verified 2013-07

CONDITIONS: Glioblastoma
Keywords: recurrent glioblastoma; multiple agents; immunotherapy; chemotherapy; brain and nervous system
MeSH Terms: conditions — Glioblastoma; Neurologic Manifestations | interventions — Vorinostat; Bevacizumab; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A - Phase I Dose Escalation (Experimental): Dose Escalation - Irinotecan and bevacizumab are given IV on days 1 and 15 of each cycle. Vorinostat is given orally on days 1-7 and 15-21 of each cycle.
  Interventions: Drug: Vorinostat; Drug: Bevacizumab; Drug: Irinotecan
- B - Treatment at Maximum Tolerated Dose (MTD) (Experimental): MTD - Treatment at maximum tolerated dose
  Interventions: Drug: Vorinostat; Drug: Bevacizumab; Drug: Irinotecan

INTERVENTIONS:
Drug: Vorinostat — Vorinostat, Bevacizumab and Irinotecan Study. Determine maximum tolerated dose for treatment.
  Other Names: NSC 701852
Drug: Bevacizumab — Vorinostat, Bevacizumab and Irinotecan Study. Determine maximum tolerated dose for treatment.
  Other Names: rhuMAb VEGF; Avastin; NSC 704865
Drug: Irinotecan — Vorinostat, Bevacizumab and Irinotecan Study. Determine maximum tolerated dose for treatment.
  Other Names: Camptosar; CPT-11; NSC 616348

SUMMARY:
The purpose of the this study is to see if an investigations cancer treatment called vorinostat can be combined with the irinotecan/bevacizumab regimen safely.

DETAILED DESCRIPTION:
Drug Administration: (A cycle is 28 days) Irinotecan and bevacizumab are given IV on days 1 and 15 of each cycle. Vorinostat is given orally on days 1-7 and 15-21 of each cycle.

Vorinostat (provided in 100mg capsules) begins at a dose of 200mg/day, escalating to 300mg/day and then to a maximum of 400mg/day. Vorinostat will be taken prior to irinotecan and bevacizumab on days 1 and 15. The drug should be administered at the same time every day for days 2-7 and 16-21. Patients will be treated prophylactically with compazine 30 minutes prior to vorinostat which, in turn, should be taken 30 minutes prior to a meal whenever possible.

Irinotecan is given at a dose of 125mg/m². Bevacizumab is given at a dose of 10mg/kg.

Maximum tolerated dose (MTD) will be defined by toxicities occurring during the first 4 weeks of therapy. Three patients will be treated at dose level one and can be enrolled simultaneously. They must be observed for dose limiting toxicities (DLT) for at least 4 weeks from treatment day 1. Page 15 of the protocol outlines the dose escalation parameters. At least 9 patients will be treated at the MTD. If DLT is not achieved in any cohort of up to a dose level of 400mg/day of vorinostat, further dose escalations will not be made. This dose will then become the recommended dose.

Patients demonstrating evidence of benefit may be treated up to a maximum of 24 cycles, at the investigator's discretion.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven intracranial glioblastoma or gliosarcoma with pathologic or radiographic confirmation of tumor progression or regrowth following standard front-line therapy. Patients will be eligible if original histology was low-grade glioma and a subsequent diagnosis of glioblastoma or gliosarcoma was made.
* History and physical examination, including neurologic examination and performance status, within 1 week prior to registration
* Systolic blood pressure ≤ 160 mmHg and diastolic pressure ≤ 90 mmHg
* Able to undergo brain magnetic resonance imaging (MRI) scans with intravenous gadolinium
* Radiographic evidence for tumor progression by MRI within 14 days prior to registration
* Karnofsky performance status ≥ 60
* Complete blood count (CBC)/differential obtained 14 days prior to registration, with adequate bone marrow function defined as follows: Absolute neutrophil count (ANC) ≥ 1,500/microL; Platelets ≥ 100,000 cells/microL; Hemoglobin ≥ 10.0 gm/dL (use of transfusion or other intervention to achieve Hgb ≥ 10.0 is acceptable)
* Adequate liver function within 14 days prior to registration, defined as follows: serum glutamic oxaloacetic transaminase (SGOT)[aspartic transaminase (AST)]/serum glutamic pyruvic transaminase (SGPT) [alanine transaminase (ALT)] < 2.5 times the upper limit of normal; Bilirubin ≤ 1.6 mg/dL
* Adequate renal function within 14 days prior to registration, defined as: Creatinine ≤ 1.5 mg/dL; Urine protein screened by urine analysis for urine protein creatinine (UPC) ratio. For UPC ratio > 0.5, 24-hour urine protein should be obtained and the level should be <1000 mg.
* If not on stable anticoagulation, prothrombin time (PT) must be within normal limits within 14 days prior to registration.
* If on full-dose anticoagulants (e.g., warfarin or LMW heparin) must meet both of the following criteria: No active bleeding or pathological condition that carries a high risk of bleeding (e.g., tumor involving major vessels or known varices); In-range international normalized ratio (INR), usually between 2 and 3) on a stable dose of oral anticoagulant or on a stable dose of low molecular weight heparin.
* Have received prior concurrent and/or adjuvant temozolomide
* Have recovered from toxic effects of prior therapy, and there must be a minimum time of 28 days from the administration of any prior cytotoxicity or investigational agent, except for nitrosureas (>42 days)
* Should not have been previously treated with any other histone deacetylase (HDAC) inhibitors (other than valproic acid for management of seizures). If they have been treated with valproic acid as treatment for seizures, the drug should be stopped at least 30 days before exposure to vorinostat.
* Should not have been previously treated with bevacizumab and/or irinotecan
* Should not have undergone more than 3 prior therapies
* Patients having undergone recent resection of recurrent or progressive tumor must meet all of the following conditions: Patients must have recovered from the effects of surgery and a minimum of 28 days must have elapsed from the day of surgery to the day of registration; If a core or needle biopsy was performed, a minimum of 7 days must have elapsed prior to registration.
* Residual disease following resection of recurrent glioblastoma is not mandated for eligibility into the study.
* Have failed prior radiation therapy and must have an interval of ≥ 42 days (6 weeks) from the completion of initial radiation therapy to registration
* Must sign study-specific informed consent prior to registration
* Women of childbearing potential (WOCBP) must have a negative β-HCG pregnancy test documented within 14 days prior to registration.
* WOCBP must agree to use 2 forms of adequate contraceptive methods. These include (1) oral, injectable, or implantable hormonal contraceptive; (2) tubal ligation; (3) intra-uterine device; (4) barrier contraceptive with spermicide; or (5) vasectomized partner. Men must also protect their partner from becoming pregnant through use of condoms with spermicide or vasectomy. Patient must agree to have standard of care MRIs.

Exclusion Criteria:

* Prior invasive malignancy that is not the glioblastoma or gliosarcoma (except nonmelanomatous skin cancer or carcinoma in situ of the cervix) unless patient has been disease free and off therapy for that disease for at least 3 years
* Acute intratumoral hemorrhage on MR imaging. Patients with MR imaging demonstrating old hemorrhage or subacute blood after a neurosurgical procedure (biopsy or resection) will be eligible for treatment.
* Must not have any significant medical illness that in the investigator's opinion cannot be adequately controlled with appropriate therapy or would compromise the patient's ability to tolerate this therapy
* Must not have any severe, active comorbidity, defined as: Transmural myocardial infarction or unstable angina within 6 months prior to study Registration; Evidence of recent myocardial infarction or ischemia by the findings of S-T elevations of ≥2 mm using the analysis of an electrocardiogram (EKG) performed within 14 days of registration; New York Heart Association (NYHA) grade II or greater or congestive heart failure requiring hospitalization within 12 months prior to registration; history of stroke or transient ischemic attack within 6 months; inadequately controlled hypertension despite antihypertensive medication; serious and inadequately controlled cardiac arrhythmia; significant vascular disease; clinically significant peripheral vascular disease; evidence of bleeding diathesis or coagulopathy; Patients on dialysis; Serious or non-healing wound, ulcer, or bone fracture; History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days prior to registration; acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration; chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within 14 days prior to registration; acquired immune deficiency syndrome (AIDS) based upon current Centers for Disease Control and Prevention (CDC); cannot be receiving highly active antiretroviral therapy (HAART); must not be diagnosed with hepatitis B or hepatitis C
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to registration
* Anticipation of need for major surgical procedures during the course of the study
* Core biopsy within 7 days prior to registration
* Pregnant or nursing breastfeeding should be discontinued prior to enrollment
* Fertile men and women who are sexually active and not willing/able to use medically acceptable forms of contraception during therapy and for at least 6 months after the completion of therapy
* Known hypersensitivity of Chinese hamster ovary cell products or other recombinant human antibodies
* Any condition that impairs ability to swallow pills
* The clearance and metabolism of irinotecan is markedly enhanced in patients receiving drugs that induce the hepatic cytochrome p450 system. In brain tumor patients, these are typically certain types of anticonvulsants, termed enzyme-inducing anti-epileptic drugs (EIAEDs). Patients cannot be receiving EIAEDs or any CYP3A4 inhibitors; patients previously receiving these agents must have discontinued their use at least 2 weeks prior to registration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2008-09; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 25 months
  Define MTD of vorinostat when combined with bevacizumab and irinotecan

SECONDARY OUTCOMES:
Number of Participants With Progression Free Survival (PFS) at 6 Months | 6 months
  All patients will be evaluable for 6 month-PFS except those that are removed from the study before the end of cycle 1 for reasons other than clinical progression (such as toxicity). Patients who suffer clinical progression without radiographic confirmation of progression will be considered to have progressive disease in determination of 6 month-PFS.
Number of Participants With Adverse Events (AEs) | 25 months
  Characterize characterize the safety profile of vorinostat in combination with bevacizumab and irinotecan. All patients will be evaluable for toxicity from the time of their first treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Prakash Chinnaiyan, M.D., Principal Investigator — H. Lee Moffitt Cancer Center & Research Institute, Inc.
Locations (1):
- H. Lee Moffitt Cancer Center & Research Institute, Inc., Tampa, Florida, United States